CLINICAL TRIAL: NCT01111799
Title: Exploration of the Possibility That Local Injury of the Endometrium Has the Same Beneficial Effect on IUI Outcome as Demonstrated in IVF Treatment
Brief Title: Does Local Injury of the Endometrium Improve Controlled Ovarian Hyperstimulation (COH) + Intrauterine Insemination (IUI) Outcome?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 004608K
Record Dates: First submitted 2010-04-21; First posted 2010-04-28 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Infertility; Implantation Failure
Keywords: endometrial biopsy; implantation; uterine receptivity; infertility; controled ovarian hyperstimulation; intra uterine insemination
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Clomiphene citrate + IUI + endometrial biopsy (Experimental): Clomiphene citrate + IUI + endometrial biopsy
  Interventions: Procedure: endometrial biopsy
- Clomiphene citrate + IUI (No Intervention)
- gonadotrophines + IUI + endometrial biopsy (Experimental): two endometrial biopsies will be taken with a PIPELLE catheter on days 12 and 21 of the spontaneous menstrual cycle that precedes the fertility treatment.
  Interventions: Procedure: endometrial biopsy
- gonadotrophines + IUI (No Intervention)
- natural cycle + IUI + endometrail biopsy (Experimental): two endometrial biopsies will be taken with a PIPELLE catheter on days 12 and 21 of the spontaneous menstrual cycle that precedes the fertility treatment.
  Interventions: Procedure: natural cycle + IUI + endometrial biopsy
- natural cycle + IUI (No Intervention)

INTERVENTIONS:
Procedure: endometrial biopsy — two endometrial biopsies will be taken with a PIPELLE catheter on days 12 and 21 of the spontaneous menstrual cycle that precedes the fertility treatment.
  Arms: Clomiphene citrate + IUI + endometrial biopsy
Procedure: endometrial biopsy — two endometrial biopsies will be taken with a PIPELLE catheter on days 12 and 21 of the spontaneous menstrual cycle that precedes the fertility treatment.
  Arms: gonadotrophines + IUI + endometrial biopsy
Procedure: natural cycle + IUI + endometrial biopsy — two endometrial biopsies will be taken with a PIPELLE catheter on days 12 and 21 of the spontaneous menstrual cycle that precedes the fertility treatment.
  Arms: natural cycle + IUI + endometrail biopsy

SUMMARY:
It was previously demonstrated in in vitro fertilization (IVF) patients that local injury of the endometrium during a spontaneous menstrual cycle that precedes IVF treatment doubled the rates of implantation and pregnancy. The hypothesis of our present study is that the endometrial injury procedure will have the same beneficial effect in patients undergoing controlled ovarian hyperstimulation (COH) combined with intrauterine insemination (IUI).

DETAILED DESCRIPTION:
In order to test our hypothesis, we will perform the simple procedure of local injury of the endometrium using a "Pipelle" biopsy catheter during the spontaneous menstrual cycle that precedes a COH + IUI treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18-38.
* infertility.
* patients undergoing IUI treatment.
* at least one failed IUI cycle.

Exclusion Criteria:

* indication for IVF treatment.
* Known Pelvic inflammatory disease(PID).

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy rate | 1 year

SECONDARY OUTCOMES:
Live birth | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Or, MD, Study Director — Clalit health service
Locations (1):
- Remez women medical center, Rehovot, Israel

REFERENCES:
- [Background] Barash A, Dekel N, Fieldust S, Segal I, Schechtman E, Granot I. Local injury to the endometrium doubles the incidence of successful pregnancies in patients undergoing in vitro fertilization. Fertil Steril. 2003 Jun;79(6):1317-22. doi: 10.1016/s0015-0282(03)00345-5. PMID 12798877